CLINICAL TRIAL: NCT05262127
Title: Clinical Assessment of the Flash Version of Eye Movement Desensitization and Reprocessing in Memory Distress: A Double Blinded Randomized Controlled Trial
Brief Title: Clinical Assessment of the Flash - Eye Movement Desensitization and Reprocessing
Acronym: Flash-EMDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Professor Kinesiology and Health Science, York University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-141
Record Dates: First submitted 2021-12-29; First posted 2022-03-02 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-02

CONDITIONS: PTSD
Keywords: behavioural internet intervention, post-traumatic stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel group, double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, assessors and care providers (if participants are in treatment) are masked to trial allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash Version of EMDR (Active Comparator): Flash methods (e.g. positive engaging focus) are used in addition to the standard EMDR techniques conveyed by video viewed online
  Interventions: Behavioral: Flash Version of EMDR
- EMDR - alone (Active Comparator): Use of standard EMDR techniques conveyed by video online
  Interventions: Behavioral: Flash Version of EMDR

INTERVENTIONS:
Behavioral: Flash Version of EMDR — EMDR and the inclusion of a positive engaging focus generated autonomously by participant

SUMMARY:
To assess the Flash version of EMDR in reductions of the disturbance of upsetting memories at post-intervention, and 1-month follow up within a double-blinded, online 2-arm randomized controlled trial (RCT) with self-report outcomes. We will assess 45 per group, adequate for the detection of a medium effect size.

This double-blinded, RCT will assess the comparative efficacy of these two online interventions designed to reduce memory disturbance.

DETAILED DESCRIPTION:
This double-blinded, RCT compares the efficacy of 2 online interventions (Flash Version - EMDR; EMDR alone) designed to reduce memory disturbance.Inclusion Criteria: (1) approved for engagement assessment by the CloudResearch platform; (2) 25-60 years; 3) US-Canada residence; (4) a recalled disturbing memory of an event that has not repeated and was moderately upsetting, or greater when event occurred; (5) memory remains moderately upsetting or greater on recall. The disturbance of upsetting memories at post-intervention, and 1-month follow up will be assessed with self-report outcomes. We will assess 45 / group, adequate for the detection of a medium effect size. linked to an earlier memory (that is equally or more disturbing). Exclusion Criteria: Diagnosis of: (1) bipolar disorder; (2) borderline personality disorder; (3) obsessive compulsive disorder; (4) schizophrenia; (5) substance abuse/addiction in the past 3 months; (6) any suicidal ideation; (7) suicide attempt in the past 6 months. Interventions: Experimental participants observe video instructions of full FT, while controls receive an online intervention that follows traditional EMDR. Measures: Primary outcome: State Anxiety subscale of the State Trait Anxiety Inventory (STAI) at baseline, post-intervention, and after 1-month follow up; Post Traumatic Stress Disorder symptoms (PTSD) measured by PCL-5 (1 month follow up).

Secondary outcomes: the Subjective Units of Disturbance (SUDs) assessing change in immediately reported disturbance of recalled memories (baseline and post-intervention); depression measured by Patient Health Questionnaire (PHQ9) and Positive-Negative Affect measured by the Positive and Negative Affect Scale (PANAS).

ELIGIBILITY:
Inclusion Criteria:

* Moderately upsetting or > memory of an event that occurred > 2 years ago and has since not repeated
* Moderately upsetting or > memory remains moderately upsetting when recalled
* Memory is not tied to an earlier memory that is equally disturbing or >

Exclusion Criteria:

* Bipolar Disorder
* Borderline Personality Disorder
* Obsessive-Compulsive Disorder
* Schizophrenia
* Substance Abuse/Addiction in past 3 months
* Suicidal ideation or attempted suicide in the past 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) 1 - 44 | 1 month follow up
  Self Report Questionnaire
State-Trait Anxiety Inventory - State 0 - 80. | 1 month follow up
  Self Report Questionnaire

SECONDARY OUTCOMES:
Patient Health Questionnaire 0 - 27 | 1 month follow up
  Self Report Questionnaire
Positive and Negative Affect Schedule 20 - 100 | 1 month followup
  Self Report Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - York University, Toronto, Ontario
  - York University - School of Kinesiology and Health Science, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Upon request, an anonymized data sheet (excel) will be sent
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 month of request
Access Criteria: Investigator at recognized academic or clinical institution

REFERENCES:
- [Derived] Babaei N, Kerry C, Goode K, Dang K, Mirzadeh P, Pirbaglou M, Kirk MA, Ritvo P. Clinical Assessment of Eye Movement Desensitization and Reprocessing in Memory Distress: Protocol for a Double-Blinded Randomized Controlled Trial. JMIR Res Protoc. 2023 May 12;12:e38552. doi: 10.2196/38552. PMID 37171869